CLINICAL TRIAL: NCT05139225
Title: A Phase Ib Study Of The Combination Of CD47 Blockade With SIRP-Alpha FC Fusion Proteins (TTI-622) And Daratumumab Hyaluronidase-fihj For Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of TTI-622 in Combination With Daratumumab Hyaluronidase-fihj in People With Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Trillium Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-122
Record Dates: First submitted 2021-10-28; First posted 2021-12-01 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: TTI-622; Daratumumab Hyaluronidase-fihj; 21-122
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: A standard 3+3 dose escalation design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TTI-622 dosing will occur over 8 weeks + Daratumumab Hyaluronidase-fihj (Experimental): TTI-622 will be administered weekly at the assigned dose levels per the ramp-up schedule. Daratumumab hyaluronidase-fihj 1800 mg will administered on a standard schedule consisting of weekly administration for 8 weeks, every other week administration for 16 weeks, followed by every 4-week administration thereafter.
  Interventions: Drug: TTI-622; Drug: Daratumumab Hyaluronidase-fihj
- TTI-622 dosing will occur over 4 weeks + Daratumumab Hyaluronidase-fihj (Experimental): TTI-622 will be administered weekly at the assigned dose levels per the ramp-up schedule. Daratumumab hyaluronidase-fihj 1800 mg will administered on a standard schedule consisting of weekly administration for 8 weeks, every other week administration for 16 weeks, followed by every 4-week administration thereafter.
  Interventions: Drug: TTI-622; Drug: Daratumumab Hyaluronidase-fihj

INTERVENTIONS:
Drug: TTI-622 — (-2) 0.4 mg/kg (-1) 0.8 mg/kg
  (1 ) 1.2 mg/kg (2) 2 mg/kg (3) 4 mg/kg (4) 8 mg/kg (5) 12 mg/kg
  The appropriate dose of TTI-622 will be administered IV over 60 minutes, however, can be extended up to 4 hours to mitigate Infusion-related reactions.
Drug: Daratumumab Hyaluronidase-fihj — Daratumumab hyaluronidase-fihj SC 1800 mg days 1, 8, 15, and 22.

SUMMARY:
This study will test the safety of TTI-622 in combination with daratumumab hyaluronidase-fihj in people with relapsed/refractory multiple myeloma. The researchers look for the highest dose TTI-622 that causes few or mild side effects in participants when given in combination with daratumumab hyaluronidase-fihj. Once the researchers find the highest safe dose of each study drug, they will further test the combination TTI-622 + daratumumab hyaluronidase-fihj) in new participants to find out if the combinations are effective in treating relapsed/refractory multiple myeloma. Researchers think that combining TTI-621 or TTI-622 with daratumumab hyaluronidase-fihj, a standard treatment for multiple myeloma, may be an effective treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory multiple myeloma, as defined by the international myeloma working group (IMWG) updated criteria (Appendix A) who have measurable disease defined by one or more of the following:

  1. Serum myeloma (M)-protein greater than or equal to 0.5 g/dL (5 g/L).
  2. Urine M-protein greater or equal to 200 mg/24 h.
  3. Involved light chain (either kappa or lambda) is >10 mg/dL with an abnormal kappa: lambda ratio.
  4. A biopsy proven plasmacytoma(s) that is new or definitely increased. Increase is defined as a 50% and at least 1 cm increase as measured serially by the sum of the products of the cross-diameters of the measurable lesion.
* Patients must have received at least 3 prior lines of therapy not having received Daratumumab Hyaluronidase-fihj in the last line of therapy, and have been previously exposed to a proteasome inhibitor, an IMiD and be considered refractory to an FD Aapproved anti-CD38 mAb used either in combination or as a single agent. Refractory is defined as progression on or within 60 days of receiving a treatment program containing an anti-CD38 monoclonal antibody.
* Female or male patients age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2. PS-3 is permitted if PS is due solely to bone pain.
* Adequate hematological function including:

  1. Absolute neutrophil count (ANC) >1,000/mm^3 (unless myelosuppression is secondary to bone marrow plasmacytosis expressed by >50% of cellularity).
  2. Platelet count >75,000/mm^3 for the dose finding portion, and > 50,000/ mm^3 for the expansion part.(transfusion is not permitted within 7 days of enrollment)
  3. Hemoglobin ≥8.0 g/dL (transfusion support is not permitted within 7 days of enrollment).
* Adequate Renal Function defined by:

  a. Estimated creatinine clearance >30 mL/min as calculated using the CKD-EPI equation. (If an estimated creatinine clearance CrCl is believed to be inaccurate for a patient, 24-hour urine collection with actual assessment of CrCl is allowed)
* Adequate Liver Function, including:

  1. Aspartate and alanine aminotransferase (AST and ALT) < 2.5 x upper limit of normal (ULN); <5.0 x ULN if there is liver involvement by the tumor.
  2. Alkaline phosphatase <2.5 x ULN (<5 x ULN in case of bone metastasis).
  3. Total bilirubin < 2.0 mg/dL, except in patients with Gilbert Syndrome who must have a total bilirubin less than 3.0 mg/dL.
* Seronegative for Hepatitis B surface (HBs) or Hepatitis B core (HBc) antigens. Patients with positive antigens must be tested for hepatitis B virus (HBV) by reverse transcription polymerase chain reaction (RT-PCR). Patients who are HBV RNA negative are eligible.
* Seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, patients must be tested for the presence of antigen by RT-PCR. Patients who are hepatitis C virus (HCV) RNA negative with adequate liver function as described above are eligible.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤ 1, with the exception of peripheral neuropathy attributable to bortezomib.
* Serum pregnancy test (for females of childbearing potential) negative at screening. Female patients of non-childbearing potential must meet at least 1 of the following criteria:

  1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state.
  2. Have undergone a documented hysterectomy and/or bilateral oophorectomy. Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.
* Signed and dated Informed Consent by study participant and/ or Legally Authorized Representative (LAR).
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures.

Exclusion Criteria:

* Patients with other malignancies in addition to multiple myeloma are not eligible if the other malignancy has required treatment within the past 3 years or is not in complete remission with the exceptions of successfully treated non-metastatic basal cell carcinoma, squamous cell skin carcinoma, or in-situ carcinoma.
* History of active autoimmune disorders (including but not limited to: Crohn's disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Grave's disease) and other conditions that require systemic therapy, which may compromise or impair the immune system.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Patients with active uncontrolled bacterial, fungal or viral infection, including known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) related illness.
* Major surgery within 4 weeks prior to study entry.
* Radiation therapy within 2 weeks prior to study entry (bone lesions requiring radiation may be treated with limited [i.e., ≤ 25% of bone marrow in field] radiation therapy during this period).
* Patients with a history of stem cell transplant (autologous or allogeneic) within 100 days prior to study enrollment.
* Donor Lymphocyte Infusion (DLI) within 30 days prior to study entry.
* Therapy with a monoclonal antibody, including but not limited to antiCD38 antibody, elotuzumab, T or NK cell re-directing therapy (ex. bispecific therapy), or antibody-drug conjugate within 30 days of study treatment initiation. Treatment with other anti-multiple myeloma therapies within 14 days of study treatment initiation.
* Patient known to be refractory to platelet or red blood cell transfusions.
* Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF, New York Heart Association Class III or IV), cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
* Fertile male patients and female patients of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Other acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 28-day observation period following C1D1 of therapy
  Dose limiting toxicities are defined as any of the following treatment emergent adverse events that occur during the 28-day DLT observation period, inclusive of pre-dose testing on C2D1. Adverse events for which a relationship to study treatment cannot be ruled out should be considered possibly related to treatment. Toxicity grading will be adjudicated according to NCI CTCAE version 5.

SECONDARY OUTCOMES:
Overall response of TTI-621 | 2 years
  measurable disease parameters and International Myeloma Working Group (IMWG) response criteria
Overall response of TTI-622 | 2 years
  measurable disease parameters and International Myeloma Working Group (IMWG) response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lesokhin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm